CLINICAL TRIAL: NCT02358057
Title: Can we Get Conscious Sedation in Optimal Safety Conditions in an Emergency Department, by Combining Dexmedetomidine With Alfentanil?
Brief Title: Can we Get Conscious Sedation by Combining Dexmedetomidine With Alfentanil?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL - DexAlf - 1
Record Dates: First submitted 2015-01-28; First posted 2015-02-06 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Procedural Sedation
Keywords: Deep sedation; Dexmedetomidine; Emergency Service, Hospital
MeSH Terms: conditions — Emergencies | interventions — Dexmedetomidine; Alfentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexmedetomidine and Alfentanil (Experimental): Patients included in the study will receive an injection of dexmedetomidine via a TIVA Injectomat Agilia, specially programmed for the injection of dexmedetomidine.
  At time zero, the patient will receive a bolus 1 mcg/ kg of dexmedetomidine during 10 minutes.
  Patients over 65 years will receive a bolus of 0.5 mcg/kg of dexmedetomidine during 10 minutes.
  Afterwards, the patient will receive a continuous injection of 0.6 mcg/kg/h of dexmedetomidine
  Patients will also receive a dose of alfentanil 1 mcg /kg, 1 minute before the technical act.
  A new alfentanil dose of 0.5 mcg / kg may be injected if pain reported by the patient corresponds to an EN > 50.
  The maximum dose of alfentanil the patient can receive is 5 mcg / kg.
  Interventions: Drug: Dexmedetomidine; Drug: Alfentanil

INTERVENTIONS:
Drug: Dexmedetomidine
  Other Names: Dexdor; Precedex
Drug: Alfentanil
  Other Names: Rapifen

SUMMARY:
The main objective is to determine if dexmedetomidine combine with alfentanil allow a level of conscious sedation within maximum security conditions in an emergency department.

Patients included in the study will receive an injection of dexmedetomidine via a TIVA Injectomat Agilia, specially programmed for the injection of dexmedetomidine.

Patients will also receive a dose of alfentanil, 1 minute before the technical act.

ELIGIBILITY:
Inclusion Criteria:

Adult over 18 years, of both sexes, for which a procedural sedation is needed in emergency room. The rules for sedation, in accordance with the international guidelines, are:

* The insertion of a chest drain
* Abscess incision and drainage
* Closed reduction of a dislocated joint

Exclusion Criteria:

* Patients refusing to participate in the study (refusal to sign the consent form)
* Patients refusing sedation
* Patients unable to participate in the study (consent is impossible to obtain)
* Pregnant women
* The hypersensitivity to the active ingredient, dexmedetomidine hydrochloride.
* Patients with poor respiratory status determined by:

Respiratory rate > 30 / min Oxygen saturation <90%

* Patients with unfavorable hemodynamic status determined by :

A heart rate > 120 / min A heart rate < 50 / min Systolic blood pressure ≥ 180 mmHg or ≤100mmHg Diastolic blood pressure ≥ 110mmHg

* Patients with contraindication to the use of dexmedetomidine :

Advanced heart block (level 2 or 3) unless pacemaker Acute cerebrovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Ramsay score scale | 2 hours

SECONDARY OUTCOMES:
Number of participants with adverse events | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Franck Verschuren, MD, PhD, Principal Investigator — St Luc